CLINICAL TRIAL: NCT01238692
Title: A Randomized Phase II Study of Oral Panobinostat (LBH589) With or Without Rituximab to Treat Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: A Phase II Study of Oral Panobinostat (LBH589) and Rituximab to Treat Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarit Assouline (Other)
Collaborators: Quebec Clinical Research Organization in Cancer (Other); Novartis (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor-Investigator, Sarit Assouline, Physician, Division of Hematology, Jewish General Hospital. Assistant Professor, Department of Oncology, McGill University, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q-CROC-02
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B cell lymphoma; DLBCL; Relapsed B-cell lymphoma; Refractory B-cell lymphoma; B-cell Lymphoma; Panobinostat; LBH589; Rituximab; Histone Deacetylase Inhibitors
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — Panobinostat; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LBH589 (Experimental)
  Interventions: Drug: LBH589
- LBH589 plus Rituximab (Experimental)
  Interventions: Drug: LBH589; Drug: Rituximab

INTERVENTIONS:
Drug: LBH589 — Patients randomized to both arms will receive oral LBH589, once-a-day, at a dose of 30 mg/day, on a three times-a-week (Monday, Wednesday and Friday) schedule as part of a 3 week (21 day) treatment cycle. Day one of each cycle will be on a Monday.
  Other Names: Panabinostat
Drug: Rituximab — Patients randomized to Arm B will receive IV rituximab at a dose of 375 mg/m2 in combination with oral LBH589. Rituximab should be administered on the same day as LBH589, after the patient has taken their LBH589 dose. The appropriate amount of solution should be withdrawn from the vial for the following calculation:
  Volume (mL) = BSA (m2) × dose (375 mg/m2) / concentration of reconstituted solution ml/mL (100 mg/10 mL and/or 500 mg/50 mL).
  Other Names: MabThera IV
  Arms: LBH589 plus Rituximab

SUMMARY:
The purpose of the study is to examine both efficacy of LBH589 in treating relapsed and refractory DLBCL, and added benefit of combining rituximab with LBH589 in this setting. Tissue samples from accessible lymph nodes will be collected and banked before the start of the study treatment and after 15 days. Additionally, blood samples will be drawn and stored in the tissue biobank.

DETAILED DESCRIPTION:
This is a randomized Phase II, multi-center study of LBH589 given alone (Arm A) or in combination with rituximab (Arm B).

The objectives of this study are:

* To investigate the efficacy of LBH589 alone and in addition to rituximab in patients with relapsed or refractory DLBCL.
* To investigate the safety and tolerability of single agent LBH589 therapy and combination therapy of LBH589 with rituximab.
* To identify potential biological factors that might correlate with efficacy.

LBH589 will be given at a dose of 30mg orally every Monday, Wednesday and Friday, as in other studies of this agent. Rituximab will be given as a single 375mg/m2 dose intravenously on day 1 of each cycle. Treatment may be administered up to 6 cycles. Treatment beyond 6 cycles will be discussed with the Sponsor. Each cycle will last 21 days.

A Phase I, dose-escalation component to the study, to determine the recommended phase II dose of rituximab in combination with LBH589, is not considered necessary as the respective toxicity profiles of these two drugs do not predict for overlapping toxicity. Dose de-escalation of LBH589 will be performed for toxicity. No dose escalations will be permitted. If patients experience grade 2 or more toxicity not returning to grade < 1 within 4 weeks after stopping therapy, they will not be allowed to continue on therapy. If more than two dose interruptions are required for toxicity, this will also be a reason to be removed from the study.

An interim analysis for safety and futility will be performed after a total of 10 patients in each arm have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of any stage of DLBCL. Patients with transformation to DLBCL will be permitted on study.
* Patients must have received at least 1 prior line of treatment if not eligible for an autologous stem cell transplant (ASCT) or 2 prior therapies, one of which must have been an ASCT, if eligible for such therapy.
* Patients must have received prior rituximab therapy and the last treatment administered with rituximab must have been given at least 6 months prior to study registration on this trial. Exception may be granted to patients treated with rituximab or other anti-CD20 monoclonal antibody 3-6 months prior to study registration upon discussion with the Sponsor.
* Patients must have at least one site of bi-dimensionally measurable lesion (> 1.5 cm in its largest dimension by CT scan).
* ECOG performance status of 0 or 1.
* Age 18 years or older.
* Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal (results 3 months prior to study registration is acceptable).
* Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.

Exclusion Criteria:

* Prior use of any anti-CD20 monoclonal antibody within 6 months of study start (refer to inclusion #3 for exception).
* History of serious infusion-related reaction to rituximab or other monoclonal antibodies.
* Central nervous system lymphoma.
* Prior treatment with HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer.
* Evidence of significant, uncontrolled concomitant disease which could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
* Impaired cardiac function
* Uncontrolled hypertension.
* Concomitant use of CYP3A4/5 inhibitors.
* Concomitant use of drugs with a risk of causing "torsades de pointes".
* Patients with unresolved diarrhea ≥ CTCAE grade 1.
* Impairment of gastrointestinal function or GI disease that may significantly alter the absorption of oral LBH589.
* Patients who have received treatment for DLBCL ≤ 3 weeks prior to starting the study treatment or who have not recovered from side effects of such therapy.
* Women who are pregnant of breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (ie. who has had menses any time preceding 12 consecutive months). WOCBP must have a negative serum pregnancy test at baseline.
* Male patients whose sexual partners are WOCBP not using double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
* Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, completely excised melanoma-in-situ, or basal or squamous cell carcinoma of the skin.
* Patients with a known positivity for HIV or hepatitis C; baseline testing for HIV and hepatitis C is not required.
* Patients with hepatitis B sAg positivity will be excluded. However, exceptions may be granted but only after discussion between the Sponsor and the site. Patients with hepatitis B core antibody positivity only must also be discussed with the Sponsor prior to entry on study (results 6 months prior to study registration is acceptable).
* Patients who cannot stop ingestion of grapefruits, starfruit, or Seville oranges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of LBH589 alone and when given in combination with rituximab | 2 years

SECONDARY OUTCOMES:
Safety and tolerability of single agent LBH589 therapy and combination therapy of LBH589 with rituximab | 2 years
Identify potential biological factors that might correlate with efficacy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Assouline, MD, Principal Investigator — Jewish General Hospital
Locations (4):
- Canada (4):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Sacré-Cœur Hospital, Montreal, Quebec

REFERENCES:
- [Result] Assouline SE, Nielsen TH, Yu S, Alcaide M, Chong L, MacDonald D, Tosikyan A, Kukreti V, Kezouh A, Petrogiannis-Haliotis T, Albuquerque M, Fornika D, Alamouti S, Froment R, Greenwood CM, Oros KK, Camglioglu E, Sharma A, Christodoulopoulos R, Rousseau C, Johnson N, Crump M, Morin RD, Mann KK. Phase 2 study of panobinostat with or without rituximab in relapsed diffuse large B-cell lymphoma. Blood. 2016 Jul 14;128(2):185-94. doi: 10.1182/blood-2016-02-699520. Epub 2016 May 10. PMID 27166360